CLINICAL TRIAL: NCT06259071
Title: Genome Wide Association Study of Patients With Muscle Specific Kinase Myasthenia Gravis
Brief Title: MuSK Myasthenia 1000 Study
Acronym: MuSK 1000
Status: Recruiting | Type: Observational
Sponsor: Myasthenia Gravis Rare Disease Network (Network)
Responsible Party: Sponsor
Other Study IDs: 8203
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Myasthenia Gravis; MuSK MG; MuSK Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MuSK myasthenia gravis 1000 study seeks to collect saliva samples from 1000 subjects with laboratory confirmed diagnosis of MuSK myasthenia to identify genetic variations associated with MuSK MG. The data collected may be used by researchers to gain a better understanding of the cause of MuSK MG and to identify biomarkers and targeted therapy for MuSK MG.

DETAILED DESCRIPTION:
Myasthenia gravis is a rare, neuromuscular (disease of the muscle and nerves) autoimmune disease characterized by weakness of the muscles. MG has a prevalence of approximately 14-40 per 100,000 people in the United States. There is no cure for MG, however understanding the disease is crucial to pave the way for development of new therapies. Important to note, the most common subtype of MG associated with Acetylcholine receptor antibodies (AChR) are found in more than 80% of patients with generalized myasthenia gravis, whereas muscle-specific kinase (MuSK) antibodies are found in only 8% of MG patients. These are found in patients with the AChR antibodies. Since the discovery of MuSK antibodies in patients, much has been learned. It has become clear that MuSK antibody MG differs in many ways from AChR antibody MG. There is some information that specific genetic factors play a role in development of MuSK MG.

Our objective is to collect saliva samples from 1000 subjects with laboratory confirmed diagnosis of MuSK myasthenia. These saliva samples will be then sent to the laboratory of Bryan Traynor who directs the Neurogenetics Laboratory at NIH. Dr. Traynor will conduct a genome-wide association study (GWAS). This study will provide important information of genetic factors leading to MuSK MG.

GWAS, also known as genome-wide association study, is a study performed to identify genetic characteristics associated with a particular disease. GWAS is currently used across various disciplines in medicine to better understand complex conditions where genetic risk factors contribute to the development of diseases.

Presently, this study has not been done in patients with MuSK MG. Researchers can use information from this study to develop quality treatment and ultimately, move toward targeted therapy approach for patients. We hope to find unique results and further enhance myasthenia research.

ELIGIBILITY:
Inclusion Criteria:

* Lab test confirming diagnosis of MuSK myasthenia gravis
* Willingness to provide saliva sample via mail or in person

Exclusion Criteria:

* Inability to provide informed consent
* Unwillingness to provide lab results of elevated muscle specific kinase antibody
* Unwillingness to provide saliva sample

Ages: 7 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: musk myasthenia gravis patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
GWAS | 2 years
  identify genetic characteristics associated with musk myasthenia gravis

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Renton AE, Pliner HA, Provenzano C, Evoli A, Ricciardi R, Nalls MA, Marangi G, Abramzon Y, Arepalli S, Chong S, Hernandez DG, Johnson JO, Bartoccioni E, Scuderi F, Maestri M, Gibbs JR, Errichiello E, Chio A, Restagno G, Sabatelli M, Macek M, Scholz SW, Corse A, Chaudhry V, Benatar M, Barohn RJ, McVey A, Pasnoor M, Dimachkie MM, Rowin J, Kissel J, Freimer M, Kaminski HJ, Sanders DB, Lipscomb B, Massey JM, Chopra M, Howard JF Jr, Koopman WJ, Nicolle MW, Pascuzzi RM, Pestronk A, Wulf C, Florence J, Blackmore D, Soloway A, Siddiqi Z, Muppidi S, Wolfe G, Richman D, Mezei MM, Jiwa T, Oger J, Drachman DB, Traynor BJ. A genome-wide association study of myasthenia gravis. JAMA Neurol. 2015 Apr;72(4):396-404. doi: 10.1001/jamaneurol.2014.4103. PMID 25643325
- [Background] Green JD, Barohn RJ, Bartoccion E, Benatar M, Blackmore D, Chaudhry V, Chopra M, Corse A, Dimachkie MM, Evoli A, Florence J, Freimer M, Howard JF, Jiwa T, Kaminski HJ, Kissel JT, Koopman WJ, Lipscomb B, Maestri M, Marino M, Massey JM, McVey A, Mezei MM, Muppidi S, Nicolle MW, Oger J, Pascuzzi RM, Pasnoor M, Pestronk A, Provenzano C, Ricciardi R, Richman DP, Rowin J, Sanders DB, Siddiqi Z, Soloway A, Wolfe GI, Wulf C, Drachman DB, Traynor BJ. Epidemiological evidence for a hereditary contribution to myasthenia gravis: a retrospective cohort study of patients from North America. BMJ Open. 2020 Sep 18;10(9):e037909. doi: 10.1136/bmjopen-2020-037909. PMID 32948566